CLINICAL TRIAL: NCT02541409
Title: Directly Observed Therapy for the Delivery of HCV Therapy Among HCV-infected Individuals in Chennai, India
Brief Title: Directly Observed Therapy for HCV in Chennai, India
Acronym: C-DOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); YR Gaitonde Centre for AIDS Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA02672; R01DA026727 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C, Chronic
Keywords: directly observed therapy; sofosbuvir; ribavirin; pegylated interferon; resource-limited setting
MeSH Terms: conditions — Hepatitis C, Chronic; Directly Observed Therapy | interventions — Sofosbuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOF+PEG+RBV (Active Comparator): Sofosbuvir (400mg/daily) + Pegylated Interferon alfa-2a (180µg/weekly) + Ribavirin (800mg/daily) for 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Pegylated Interferon alfa-2a; Drug: Ribavirin
- SOF+RBV (Active Comparator): Sofosbuvir (400mg/daily) + Ribavirin (800mg/daily) for 24 weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — Direct acting antiviral agent used for the treatment of hepatitis C
  Other Names: Sovaldi, Hepcvir, MyHep, Hepcinat, Resof, SoviHep
Drug: Pegylated Interferon alfa-2a — Antiviral agent used for the treatment of hepatitis C
  Other Names: Pegasys, Taspiance
  Arms: SOF+PEG+RBV
Drug: Ribavirin — Antiviral agent (guanosine analogue) used for the treatment of hepatitis C
  Other Names: Rebetol, Copegus, Univirin

SUMMARY:
The primary objective of this pilot trial is to evaluate the feasibility of 12 weeks vs. 24 weeks of field-based directly observed therapy (DOT) for HCV therapy in a resource-limited setting. The investigators will compare treatment completion rates among 50 persons chronically infected with HCV who will be randomized to receive either 1) 12 weeks of sofosbuvir (SOF) + ribavirin (RBV) + pegylated interferon alfa-2a (PEG); or 2) 24 weeks of SOF + RBV. Treatment will be delivered daily by field workers at a location of a participants choosing. Secondary objectives are 1) To compare the efficacy of SOF+RBV with or without PEG as measured by the proportion of subjects with sustained viral response at 12 weeks after discontinuation of therapy (SVR12); 2) To evaluate the safety and tolerability of SOF+RBV with or without PEG; 3) To assess the impact of SVR12 on insulin resistance.

DETAILED DESCRIPTION:
This will be a non-blinded randomized clinical trial with 50 participants randomized at a 1:1 allocation ratio to one of two treatment arms.

Arm 1: Sofosbuvir (400mg/daily) + Pegylated Interferon alfa-2a (180µg/weekly) + Ribavirin (800mg/daily) for 12 weeks

Arm 2: Sofosbuvir (400mg/daily) + Ribavirin (800mg/daily) for 24 weeks

Pegylated-interferon alfa-2a (PEG) will be delivered subcutaneously once weekly. Sofosbuvir (SOF) and ribavirin (RBV) will be taken orally once daily for the entire study period.

The study will take place at the YR Gaitonde Centre for AIDS Research and Education (YRGCARE). YRG CARE is a non-profit medical and research institution in Chennai. YRGCARE Medical Centre provides medical care for more than 18,000 persons with HIV disease. Currently more than 8000 persons are receiving highly active antiretroviral therapy at the center.

Participants will be recruited from the YR Gaitonde Centre for Substance Abuse Research (YRGCSAR), which is affiliated with YRGCARE. The investigators will primarily recruit subjects from a cohort study of current and former people who inject drugs (PWID) that is ongoing at the same center. Eligible participants will be randomized to one of the two treatment arms after providing written informed consent. Treatment will be delivered directly to participants daily by field workers at a location of the participants choosing. Participants will be asked to visit the study clinic every four weeks during treatment and 12 weeks after completing treatment for additional study procedures. In addition, participants in Arm 1 will be asked to visit the clinic every week to receive their PEG injection.

The primary outcome is treatment completion. Secondary outcomes include SVR12, safety and tolerability and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Willing/able to provide consent
2. Age ≥ 18
3. Chronic HCV (HCV RNA positive)
4. Resident of Chennai and can provide locator information
5. If co-infected with HIV, must have CD4 (Cluster of Differentation 4) > 350 cells/mm3 and either: 1) ART naïve or 2) if on ART be on a tenofovir-containing regimen. If a participant's CD4 drops below 350 cells/μl (threshold for treatment in India), will have to initiate a tenofovir-containing regimen (current standard of care).
6. Participants must have the following at screening:

   1. Alanine Aminotransferase (ALT) ≤ 10 x the upper limit of normal (ULN)
   2. Aspartate Aminotransferase (AST) ≤ 10 x ULN
   3. Hemoglobin ≥ 12 g/dl for males and 11 g/dl for females
   4. International normalized ratio (INR) ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   5. Albumin ≥ 3 g/dl
   6. Direct bilirubin ≤ 1.5 x ULN
   7. Creatinine clearance ≥ 60 ml/min (Cockgroft-Gault Equation)
   8. Alpha fetoprotein < 50 ng/ml
   9. Absolute neutrophil count (ANC) ≥ 1,500/μL
   10. Platelets ≥ 90,000/μL
   11. Thyroid stimulating hormone (TSH) ≤ ULN
7. A female subject is eligible if it is confirmed that she is:

   1. Not pregnant or nursing
   2. Of non-childbearing potential (i.e., women who have had hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation (for ≥12 months) of previously occurring menses
   3. Of childbearing potential and negative urine pregnancy test prior to randomization and agree to one of the following from 3 weeks prior to Baseline/Day 1 until 6 months after the last dose of RBV.

      * Complete abstinence from intercourse.

   Or

   • Consistent use of approved methods of birth control in addition to a male partner who correctly uses a condom from 3 weeks prior to Baseline/Day 1 until 6 months after the last dose of RBV.
8. Male participants must agree to consistently and correctly use a condom. If their female partner is of childbearing potential, their partner must agree to use one of the study approved non-hormonal methods of birth control or a hormone-containing contraceptive, from the date of screening until 7 months after their last dose of RBV
9. Male participants must agree to refrain from sperm donation for at least 7 months after the last dose of RBV.
10. Of generally good health as determined by the investigator.
11. Able to comply with the dosing instructions for study drug administration and willing to complete the study schedule of assessments.

Exclusion Criteria:

1. Pregnant/nursing female or male with pregnant/nursing female partner.
2. Current or prior history of clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage, MELD<12)
3. Prior hepatitis C treatment
4. Infection with hepatitis B virus
5. Chronic use of systematically administered immunosuppressive agents (e.g., prednisone equivalent >10 mg/day)
6. Use of any prohibited concomitant medications within 28 days of the Baseline/Day 1 visit.
7. Contraindications to RBV therapy or PEG/RBV
8. Known hypersensitivity to RBV or PEG, the metabolites or formulation excipients
9. Additional exclusion criteria related to Aim 1 regimen

   1. Pre-existing significant psychiatric condition(s) including severe depression, severe bipolar disorder and schizophrenia. Other psychiatric disorders are permitted if the condition is well controlled with a stable treatment regimen for ≥ 1 year from screening.
   2. Presence of autoimmune disorders (e.g., systemic lupus erythematosus, rheumatoid arthritis, sarcoidosis).
   3. History of clinical significant retinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil S Solomon, MBBS, PhD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- YR Gaitonde Centre for AIDS Research and Education, Chennai, Tamil Nadu, India

REFERENCES:
- [Derived] Solomon SS, Sulkowski MS, Amrose P, Srikrishnan AK, McFall AM, Ramasamy B, Kumar MS, Anand S, Thomas DL, Mehta SH. Directly observed therapy of sofosbuvir/ribavirin +/- peginterferon with minimal monitoring for the treatment of chronic hepatitis C in people with a history of drug use in Chennai, India (C-DOT). J Viral Hepat. 2018 Jan;25(1):37-46. doi: 10.1111/jvh.12761. Epub 2017 Aug 14. PMID 28719029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOF+PEG+RBV | SOF+RBV
Started | 25 | 25
Completed | 22 | 22
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOF+PEG+RBV | SOF+RBV | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [41 to 50] | 46 [44 to 47] | 46 [42 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 25 | 25 | 50
HCV Genotype 3a [Count of Participants; unit: Participants] | 22 | 20 | 42
HCV Genotype 1a [Count of Participants; unit: Participants] | 2 | 5 | 7
HCV Genotype 6n [Count of Participants; unit: Participants] | 1 | 0 | 1
Lifetime Injection Drug Use: Heroin [Count of Participants; unit: Participants] | 24 | 25 | 49
Lifetime Injection Drug Use: Sedatives [Count of Participants; unit: Participants] | 19 | 16 | 35
Lifetime Injection Drug Use: Other Opioids [Count of Participants; unit: Participants] | 24 | 23 | 47
Injection Drug use in Prior 6 Months [Count of Participants; unit: Participants] | 1 | 0 | 1
NonInjection Drug Use in Prior 6 Months [Count of Participants; unit: Participants] | 7 | 2 | 9
Marijuana Use in Prior 6 Months [Count of Participants; unit: Participants] | 4 | 1 | 5
No Alcohol Use in Prior 6 Months [Count of Participants; unit: Participants] | 14 | 13 | 27
Alcohol Use in Prior 6 Months: 1-4 Drinks Daily [Count of Participants; unit: Participants] | 9 | 9 | 18
Alcohol Use in Prior 6 Months: >5 Drinks Daily [Count of Participants; unit: Participants] | 2 | 3 | 5
Alcohol Use: No/Mild Alcohol Use [Count of Participants; unit: Participants] | 14 | 14 | 28
Alcohol Use: Harmful/Hazardous Alcohol Use [Count of Participants; unit: Participants] | 1 | 2 | 3
Alcohol Use: Alcohol Dependence [Count of Participants; unit: Participants] | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: HCV Treatment Completion
Description: The percentage of subjects that complete their course of treatment
Time Frame: 12 weeks from baseline for SOF+PEG+RBV and 24 weeks from baselne for SOF+RBV
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+PEG+RBV | SOF+RBV
Number analyzed (Participants) | 25 | 25
Participants | 22 | 22

2. Secondary Outcome: Sustained Virologic Response (SVR)
Description: The percentage of participants who achieve SVR as assessed by undetectable HCV RNA measured 12 weeks after treatment completion
Time Frame: 24 weeks from baseline for SOF+PEG+RBV and 36 weeks from baseline for SOF+RBV
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+PEG+RBV | SOF+RBV
Number analyzed (Participants) | 25 | 25
Participants | 22 | 15

3. Secondary Outcome: Serious Adverse Events
Description: Number of participants with treatment-related serious adverse events by laboratory tests and physician examination
Time Frame: 24 weeks from baseline SOF+PEG+RBV and 36 weeks from baseline for SOF+RBV
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+PEG+RBV | SOF+RBV
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

4. Secondary Outcome: Change in Insulin Resistance
Description: Change in insulin resistance while on treatment by the homeostasis model assessment - insulin resistance (HOMA-IR). HOMA-IR is calculated according to the formula (fasting insulin (microU/L)+fasting glucose (nmol/L)/22.5. Fasting insulin and glucose measurements are obtained using whole blood.
Time Frame: Difference from entry to 24 weeks for SOF+PEG+RBV and difference from entry to 36 weeks for SOF+RBV
Measure: Median (Inter-Quartile Range); unit: HOMA-IR
Arm/Group | SOF+PEG+RBV | SOF+RBV
Number analyzed (Participants) | 25 | 25
HOMA-IR | 1.2 [-0.1 to 9.1] | 0.2 [-1.3 to 6.0]

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | SOF+PEG+RBV | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No